CLINICAL TRIAL: NCT06663020
Title: Impact of Smoking Cessation Duration on Postoperative Complications in Lung Cancer Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Caner İşevi, MD (Other)
Responsible Party: Sponsor-Investigator, Caner İşevi, MD, Thoracic Surgeon, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Other Study IDs: B.30.2.ODM.0.20.08/19
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2024-12

CONDITIONS: Smoking Cessation; Lung Cancer (NSCLC); Postoperative Complication
Keywords: lung cancer; smoking cessation; postoperative complication; thoracic surgery
MeSH Terms: conditions — Smoking Cessation; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Smoking Cessation Duration — Participants are categorized based on their smoking status and the duration since they quit smoking prior to lung cancer surgery. This observational study focuses on evaluating the relationship between the duration of smoking cessation (measured in days or weeks) and the incidence of postoperative complications. Smoking cessation duration is recorded for each participant to determine its impact on surgical outcomes.

SUMMARY:
This study aims to investigate the relationship between the duration of smoking cessation before surgery and postoperative complications in lung cancer patients undergoing surgery. Lung cancer surgery patients who have recently quit smoking or are long-term nonsmokers will be evaluated to determine if the timing of smoking cessation impacts the risk of complications after surgery. By analyzing these factors, the study seeks to provide guidance on optimal smoking cessation timing to reduce postoperative risks.

DETAILED DESCRIPTION:
This prospective observational study aims to examine the impact of smoking cessation duration on postoperative complications in lung cancer surgery patients. Lung cancer remains the most lethal type of cancer globally, with non-small cell lung cancer (NSCLC) accounting for approximately 85% of cases. Tobacco use is the most well-established risk factor for lung cancer, and a significant portion of lung cancer patients have either smoked in the past or continue to smoke. Smoking status and the timing of cessation before surgery have been shown to influence postoperative outcomes. Prior research suggests that cessation at least 2-4 weeks before surgery may reduce postoperative complications, with the World Health Organization recommending a minimum of four weeks of cessation before surgery to decrease the risk of adverse outcomes.

In this study, patients will not be categorized based on smoking or cessation status alone but will be documented on a continuum by recording the exact number of days or weeks between their smoking cessation and their surgical procedure. The primary objective is to assess whether a specific duration of smoking cessation is associated with a reduced risk of postoperative complications, including both pulmonary and non-pulmonary complications. These complications are defined in two categories: respiratory (e.g., atelectasis, pneumonia, respiratory failure) and non-respiratory (e.g., atrial fibrillation, myocardial infarction, wound infection).

Patients with advanced chronic obstructive pulmonary disease (COPD), uncontrolled asthma, severe neuromuscular disease, advanced thoracic deformity, or severe cardiovascular disease will be excluded to minimize confounding variables. The study will also exclude patients with emergency surgeries, pregnant individuals, and those who have undergone prior thoracic surgeries.

The sample size calculation, performed using G*Power software, determined a minimum of 248 participants would be needed to achieve a 95% confidence level and statistical power of 95%. Data analysis will include logistic regression to examine the relationship between smoking cessation duration and the occurrence of postoperative complications. Risk assessment tools, including the ARISCAT, Gupta Postoperative Pneumonia Risk, and Melbourne Group Scale, will be utilized to evaluate each patient's risk profile.

Data collection will focus on the following variables:

Patient demographics, comorbidities, neoadjuvant therapy, preoperative smoking history, lung function tests, operative and anesthesia times, intraoperative blood loss, pathological staging, and 30-day postoperative complications.

Quality assurance will involve source data verification from medical records to ensure accuracy, as well as routine data validation checks to maintain data consistency.

The statistical analysis will be guided by a comprehensive analysis plan, detailing the primary and secondary outcome evaluations. The findings aim to contribute to understanding the optimal smoking cessation timing to reduce surgical risks and enhance patient outcomes in lung cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80 years.
* Patients scheduled for elective surgery under general anesthesia due to NSCL.
* Patients classified as American Society of Anesthesiologists (ASA) I-III.
* Patients or their legally authorized representatives who have provided informed consent.

Exclusion Criteria:

* Patients with advanced chronic obstructive pulmonary disease (COPD) classified as GOLD Grade III-IV.
* Patients with severe and uncontrolled bronchial asthma.
* Patients with severe neuromuscular diseases or advanced thoracic deformity.
* Patients with severe heart disease classified as New York Heart Association (NYHA) Class III-IV.
* Patients with cognitive impairments.
* Patients undergoing emergency surgery.
* Pregnant patients.
* Patients with coagulopathy.
* Patients who have previously undergone video-assisted thoracoscopic surgery (VATS) and/or thoracotomy.
* Patients who died perioperatively.
* Patients or their legally authorized representatives who did not provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from patients diagnosed with non-small cell lung cancer at the Ondokuz Mayis University Medical Faculty, Department of Thoracic Surgery. The study population consists of individuals scheduled for elective lung cancer surgery under general anesthesia, reflecting a clinical sample of patients who are typically managed within a tertiary care hospital setting.
Sampling Method: Non-Probability Sample
Enrollment: 248 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Complications Among Patients Following Lung Cancer Surgery Based on Duration of Smoking Cessation | From the day of surgery to 30 days postoperatively
  Postoperative complications will be assessed in patients who have undergone lung cancer surgery. Complications include both pulmonary (e.g., pneumonia, atelectasis, prolonged air leak) and non-pulmonary events (e.g., atrial fibrillation, wound infection) occurring within 30 days after surgery. The duration of smoking cessation prior to surgery will be recorded for each patient, and complications will be documented according to standard clinical criteria. This measure aims to determine if the length of smoking cessation impacts the likelihood and type of postoperative complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University Medical Faculty, Department of Thoracic Surgery, Samsun, Samsun, Turkey (Türkiye)